CLINICAL TRIAL: NCT06409676
Title: Applicability of Enhanced Recovery After Surgery Protocols in the Therapeutic Endoscopy Suite: a Single-Center Randomized Prospective Study
Brief Title: Applicability of Enhanced Recovery After Surgery Protocols in the Therapeutic Endoscopy Suite
Acronym: ERATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ERATE ID. 3764
Record Dates: First submitted 2024-02-16; First posted 2024-05-10 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Endoscopic Submucosal Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS group (Experimental): Participants will receive the ERAS protocol tailored for endoscopic procedures
  Interventions: Procedure: ERAS protocols
- Standard care group (No Intervention): Participants will receive conventional pre-endoscopic care, including basic patient education, standard bowel preparation, preoperative fasting guidelines, medication management, and routine preoperative assessment

INTERVENTIONS:
Procedure: ERAS protocols — Enhanced Recovery After Surgery (ERAS) guidelines are evidence-based recommendations aimed at improving patient outcomes and reducing complications after surgery.
  Arms: ERAS group

SUMMARY:
This study aims to investigate the impact of implementing ERAS protocols on patient outcomes in therapeutic endoscopy, focusing on patients undergoing ESD. Although considered a less invasive alternative to conventional surgical resection, ESD can still result in significant physiological stress, postoperative discomfort, and potential complications. By exploring the application of ERAS principles to therapeutic endoscopy and evaluating their effectiveness, this study aims to address the current lack of knowledge in this field and promote the adoption of ERAS principles in managing ESD patients. Ultimately, the goal is to assess if the implementation of the ERAS process in these therapeutic endoscopy procedures can reduce procedure-related complications, improve patient outcomes, and enhance after-procedural recovery.

ELIGIBILITY:
Inclusion Criteria:

* All >18 years-old patients scheduled for ESD for any indication;
* Patients who were able to give informed written consent.

Exclusion Criteria:

* - Patients who were not able or refused to give informed written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of ESD-related adverse events | 48 hours after procedure
  such as bleeding or perforation (defined as any such procedure-related complication that compromises the completeness of the procedure and/or results in the unplanned patient hospital admission) or occurrence of Post Endoscopic submucosal dissection Coagulation Syndrome (PECS).
  (defined as the presence of signs of inflammation, such as fever, leukocytosis or C-reactive protein in the presence of localized abdominal pain in patients without evidence of perforation to
airway protection | during procedure
  Desaturations, aspiration or any acute event requiring airway protection

SECONDARY OUTCOMES:
Post-procedural Recovery | 24-48 hours after procedure
  Assessed using the Postoperative Quality of Recovery Scale (PQRS)
Overall patient satisfaction | 24-48 hours after procedure
  which will be evaluated using a 0-10 scale (0 = highly unsatisfactory outcome, 10 = most satisfactory outcome) or the Patient Satisfaction Questionnaire-18 (PSQ-18))
Abdominal pain | at 3 and 6 hours after endoscopy
  which will be assessed using the NRS (with a range from 0 to 10, where 0 corresponds to no pain while 10 to the worst pain imaginable)
Analgesic requirements | in the 24 hours after ESD
  which will be assessed using the NRS (with a range from 0 to 10, where 0 corresponds to no pain while 10 to the worst pain imaginable )
PADSS: Post Anesthetic Discharge Scoring System (evaluated from 0 to 2, using: Vital signs, Activity and mental status, Pain, nausea and/or vomiting, Surgical bleeding, Intake and output) | in the first 4 hours after ESD
  % of patients with PADSS >=9

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ficari F, Borghi F, Catarci M, Scatizzi M, Alagna V, Bachini I, Baldazzi G, Bardi U, Benedetti M, Beretta L, Bertocchi E, Caliendo D, Campagnacci R, Cardinali A, Carlini M, Cascella M, Cassini D, Ciotti S, Cirio A, Coata P, Conti D, DelRio P, Di Marco C, Ferla L, Fiorindi C, Garulli G, Genzano C, Guercioni G, Marra B, Maurizi A, Monzani R, Pace U, Pandolfini L, Parisi A, Pavanello M, Pecorelli N, Pellegrino L, Persiani R, Pirozzi F, Pirrera B, Rizzo A, Rolfo M, Romagnoli S, Ruffo G, Sciuto A, Marini P. Enhanced recovery pathways in colorectal surgery: a consensus paper by the Associazione Chirurghi Ospedalieri Italiani (ACOI) and the PeriOperative Italian Society (POIS). G Chir. 2019 Jul-Aug;40(4Supp.):1-40. PMID 32003714
- [Background] Ahmed J, Khan S, Lim M, Chandrasekaran TV, MacFie J. Enhanced recovery after surgery protocols - compliance and variations in practice during routine colorectal surgery. Colorectal Dis. 2012 Sep;14(9):1045-51. doi: 10.1111/j.1463-1318.2011.02856.x. PMID 21985180
- [Background] Wang Y, Zhu Z, Li H, Sun Y, Xie G, Cheng B, Ji F, Fang X. Effects of preoperative oral carbohydrates on patients undergoing ESD surgery under general anesthesia: A randomized control study. Medicine (Baltimore). 2019 May;98(20):e15669. doi: 10.1097/MD.0000000000015669. PMID 31096498
- [Background] Li J, Kang G, Liu T, Liu Z, Guo T. Feasibility of Enhanced Recovery After Surgery Protocols Implemented Perioperatively in Endoscopic Submucosal Dissection for Early Gastric Cancer: A Single-Center Retrospective Study. J Laparoendosc Adv Surg Tech A. 2023 Jan;33(1):74-80. doi: 10.1089/lap.2022.0269. Epub 2022 Jun 20. PMID 35723625
- [Background] Wang Y, Zhou D, Xiong W, Ge S. Modified protocol for Enhanced Recovery After Surgery is beneficial for achalasia patients undergoing peroral endoscopic myotomy: a randomized prospective trial. Wideochir Inne Tech Maloinwazyjne. 2021 Dec;16(4):656-663. doi: 10.5114/wiitm.2021.104013. Epub 2021 Mar 1. PMID 34950259
- [Background] Greco M, Capretti G, Beretta L, Gemma M, Pecorelli N, Braga M. Enhanced recovery program in colorectal surgery: a meta-analysis of randomized controlled trials. World J Surg. 2014 Jun;38(6):1531-41. doi: 10.1007/s00268-013-2416-8. PMID 24368573
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- [Background] ASGE Standards of Practice Committee; Early DS, Lightdale JR, Vargo JJ 2nd, Acosta RD, Chandrasekhara V, Chathadi KV, Evans JA, Fisher DA, Fonkalsrud L, Hwang JH, Khashab MA, Muthusamy VR, Pasha SF, Saltzman JR, Shergill AK, Cash BD, DeWitt JM. Guidelines for sedation and anesthesia in GI endoscopy. Gastrointest Endosc. 2018 Feb;87(2):327-337. doi: 10.1016/j.gie.2017.07.018. Epub 2018 Jan 3. No abstract available. PMID 29306520
- [Background] Jin S, Liang DD, Chen C, Zhang M, Wang J. Dexmedetomidine prevent postoperative nausea and vomiting on patients during general anesthesia: A PRISMA-compliant meta analysis of randomized controlled trials. Medicine (Baltimore). 2017 Jan;96(1):e5770. doi: 10.1097/MD.0000000000005770. PMID 28072722
- [Background] Skolnik A, Gan TJ. Update on the management of postoperative nausea and vomiting. Curr Opin Anaesthesiol. 2014 Dec;27(6):605-9. doi: 10.1097/ACO.0000000000000128. PMID 25225824
- [Background] Chen HY, Deng F, Tang SH, Liu W, Yang H, Song JC. Effect of different doses of dexmedetomidine on the median effective concentration of propofol during gastrointestinal endoscopy: a randomized controlled trial. Br J Clin Pharmacol. 2023 Jun;89(6):1799-1808. doi: 10.1111/bcp.15647. Epub 2023 Jan 9. PMID 36527308